CLINICAL TRIAL: NCT05537714
Title: Advancing Vaccine Equity: A Mixed-methods Study to Understand Vaccine Hesitancy, Structural Barriers, and Trust in Vaccine Information Among Medically Underserved Populations Living in the Rural South
Brief Title: Advancing Vaccine Equity Through Understanding Vaccine Hesitancy, Barriers, and Trust
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: East Carolina University (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0682
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Vaccine Hesitancy; Structural Barriers; Vaccine Trust
MeSH Terms: conditions — Vaccination Hesitancy | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaccine hesitant: We will conduct quantitative (survey) and qualitative assessments (interviews/focus groups) with 40 vaccine hesitant, Black, Hispanic, and medical underserved individuals living in rural eastern North Carolina (ENC)
  Interventions: Behavioral: Qualitative interviews/focus groups
- Trusted community leaders: We will conduct quantitative (survey) and qualitative assessments (interviews/focus groups) with 40 trusted individuals such as clergy/church leaders, community health workers, and community leaders who serve medical underserved individuals living in rural eastern North Carolina (ENC) .
  Interventions: Behavioral: Qualitative interviews/focus groups

INTERVENTIONS:
Behavioral: Qualitative interviews/focus groups — We will conduct quantitative (survey) and qualitative assessments (interviews/focus groups) with 40 vaccine hesitant, Black, Hispanic, and medical underserved individuals living in rural eastern North Carolina (ENC) and with 40 trusted individuals such as clergy/church leaders, community health workers, and community leaders who serve these populations.

SUMMARY:
In the proposed study, the investigators will conduct qualitative interviews and focus groups with Black, Hispanic, and medically underserved communities, living in the rural south and will provide a quantitative survey (mixed methods) to identify reasons for vaccine hesitancy, including any structural barriers experienced by this population. The investigators will assess what vaccination messaging was received by trusted individuals and how this messaging may have impacted vaccination behavior. This mixed methods study design will allow for a comprehensive picture of vaccine equity and hesitancy for this population. The quantitative survey provides a focused and concrete uncovering of the issues and relationships and the qualitative design allows for a detailed, contextualized insight into lived experiences. Coupled together, this mixed methods design will provide a rich depiction of the underlying drivers of vaccine hesitancy, structural barriers to vaccination, and messaging that impacted uptake for medically underserved and rural populations.

DETAILED DESCRIPTION:
Objective 1: To identify reasons for vaccine hesitancy, structural barriers to vaccination, vaccine messaging received, and vaccination behavior among medically underserved and vulnerable populations living in the rural south.

Objective 2: To assess vaccine messaging from trusted individuals (e.g., clergy/church leaders, community health workers, and community leaders) who serve medically underserved and vulnerable populations living in the rural south.

Objective 3: To identify best vaccine confidence and uptake strategies to improve vaccine acceptance, confidence, and trust among medically underserved and vulnerable populations living in the rural south.

Hypotheses:

H1a. It is hypothesized that top reasons for vaccine hesitancy may include access to care issues (such as transportation, long wait times, no available appointments, not sure where to go, no internet, and language barriers), safety and efficacy concerns, distrust in government and health organizations, as well as lack of information and/or misinformation.

H1b. It is hypothesized that structural barriers to vaccination may include geographic barriers, access to information, clinic/outlet location or trusted points of access, internet access, immigrant status, language, transportation, among others.

H1c. It is hypothesized that vaccine messaging received from trusted individuals in the communities (i.e., faith-based leaders, community health workers, and community leaders) will have impacted confidence and uptake more so than other vaccine messaging efforts.

H2. It is hypothesized that the vaccine messaging from trusted individuals will be mixed with some messaging based on science and some based on anecdotal evidence. It is not well-known what messages are being delivered around vaccination from trusted individuals who serve our priority population and thus, we can only hypothesize that the messaging will vary.

H3. It is hypothesized that the most effective strategies to boost vaccine confidence and uptake for vaccine hesitant, medically underserved, and vulnerable populations living in the rural south will include culturally tailored messaging from engagement with trusted individuals.

ELIGIBILITY:
Inclusion Criteria: All English or Spanish speaking adults 18 years or older. -

Exclusion Criteria: Anyone over 18 years of age who does not speak English or Spanish or anyone under 18 years of age.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eastern North Carolina (ENC) is a largely rural, poor, and underserved region of the state with 1 in 5 adults living below the poverty level, and nearly half living in a community designated as rural. Health in ENC is significantly poorer than health in the rest of NC, and health in the ENC-29 counties is poorest of all. Of the 40 counties in NC that are most economically distressed, 19 (48%) are in the ENC-29-county sub- region. Residents of ENC experience a high burden of health disparities driven by limited access to healthcare and inequitable distribution of social determinants of health.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-08-06 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Perceptions of community members | 2 years
  Topical guide questions for community members will include questions regarding vaccine hesitancy, barriers experienced to vaccination, vaccine messaging likes and dislikes, trust in vaccine message deliverers, and vaccination behavior for self and children.
Perceptions of community leaders | 2 years
  Topical guide questions for trusted individuals will include questions regarding vaccine hesitancy of themselves, vaccine hesitancy of the populations they serve, perceived barriers to vaccination of those they serve, vaccine beliefs and attitudes, trust in vaccine messaging delivered from government/healthcare system, and experience in delivering vaccine messaging to the populations they serve.

CONTACTS AND LOCATIONS:
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data can be shared upon reasonable request.